CLINICAL TRIAL: NCT00112671
Title: A Phase II Study of BAY 43-9006 in Advanced or Metastatic Urothelial Cancer (Transitional Cell Cancer of the Bladder, Ureter and Renal Pelvis)
Brief Title: Sorafenib in Treating Patients With Advanced or Metastatic Cancer of the Urinary Tract
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03095; PHL-036; 7062; N01CM62203 (NIH)
Record Dates: First submitted 2005-06-02; First posted 2005-06-03 (Estimated); Results first posted 2015-09-03 (Estimated); Last update posted 2018-07-27 (Actual); Status verified 2018-07

CONDITIONS: Metastatic Transitional Cell Cancer of the Renal Pelvis and Ureter; Recurrent Bladder Cancer; Recurrent Transitional Cell Cancer of the Renal Pelvis and Ureter; Regional Transitional Cell Cancer of the Renal Pelvis and Ureter; Stage III Bladder Cancer; Stage IV Bladder Cancer; Transitional Cell Carcinoma of the Bladder
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Sorafenib

ARMS (1):
- Treatment (sorafenib tosylate) (Experimental): Patients receive oral sorafenib twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: sorafenib tosylate; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: sorafenib tosylate — Given orally 400mg orally twice daily
  Other Names: BAY 43-9006; BAY 43-9006 Tosylate Salt; BAY 54-9085; Nexavar; SFN
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying how well sorafenib works in treating patients with advanced or metastatic cancer of the urinary tract. Sorafenib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the efficacy (response rate and stable disease rate) of Bay 439006 given to patients with advanced or metastatic urothelial cancer.

II. To assess the toxicity, time to progression and response duration of Bay 439006 given to patients with advanced or metastatic urothelial cancer.

III. To measure Ras mutational status and EGFR/HER2 on archival specimens. To determine baseline and post-treatment levels of pERK, pAKT, VEGFR2, CD31, Ki-67/MIB-1, and cleaved caspase 3 and to explore the relationship between these correlative endpoints and clinical outcome.

OUTLINE: This is a nonrandomized, open-label, multicenter study.

Patients receive oral sorafenib twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed within 3 weeks and then every 3 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed transitional cell cancer of the bladder, renal pelvis or ureter
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 20 mm with conventional techniques or as >= 10 mm with spiral CT scan
* Patients must not have had any prior systemic therapy for advanced or metastatic disease; prior adjuvant or neoadjuvant chemotherapy is permitted providing it was completed at least 4 weeks prior to study entry; radiation therapy is permitted if completed > 4 weeks prior to trial entry
* Life expectancy of greater than 3 months
* ECOG performance status 0 or 1 (Karnofsky >= 70%)
* Leukocytes >= 3,000/uL
* Absolute neutrophil count >= 1,500/uL
* Platelets >= 100,000/uL
* Total bilirubin within normal institutional limits
* AST(SGOT)/ALT(SGPT) =< 2.5 X institutional upper limit of normal
* Creatinine < 1.5 x ULN OR creatinine clearance >= 45 mL/min/1.73 m^2
* No serious medical conditions such as myocardial infarction within 6 months prior to entry, congestive heart failure, unstable angina, active cardiomyopathy, unstable ventricular arrhythmia, uncontrolled hypertension, uncontrolled psychotic disorders, serious infections, active peptic ulcer disease, or any other medical conditions that might be aggravated by treatment
* Patients must have tumor lesions accessible for biopsy for correlative studies and must be willing to undergo tumor biopsy once before and once during experimental therapy; if there is a medical contraindication to biopsy, exception may be granted upon discussion with the Principal Investigator/Chair
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Able to swallow and retain oral medication
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Prior systemic therapy for advanced or metastatic urothelial carcinoma
* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents
* Patients receiving any other investigational agents, or concurrent anticancer therapy
* Patients with only non-measurable disease, defined as all other lesions, including small lesions (longest diameter < 20mm with conventional techniques or < 10 mm with spiral CT scan) and truly non-measurable lesions, which include the following:

  * Bone lesions
  * Leptomeningeal disease
  * Ascites
  * Pleural/pericardial effusion
  * Inflammatory breast disease
  * Lymphangitis cutis/pulmonis
  * Abdominal masses that are not confirmed and followed by imaging techniques
  * Cystic lesions
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound evaluation of neurologic and other adverse events
* Patients with a history of other active malignancy in the past 5 years (with the exception of adequately treated cervical carcinoma in situ and non melanomatous skin cancers) are excluded
* Uncontrolled intercurrent illness including, but no limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients must not have any evidence of a bleeding diathesis
* Patients must not be on therapeutic anticoagulation; prophylactic anticoagulation (ie. Low dose warfarin) of venous or arterial access devices is allowed provided that the requirements for PT, INR or PTT are met
* Patients must not be taking the cytochrome P450 enzyme-inducing antiepileptic drugs (phenytoin, carbamazepine, or Phenobarbital), rifampin or St. John's Wort
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with BAY 43-9006
* Patients with immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy; therefore, HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to BAY 43-9006
* Patients with GI tract disease resulting in an inability to take oral medication, malabsorption syndrome, a requirement for IV alimentation, prior surgical procedures affecting absorption, uncontrolled inflammatory GI disease (e.g., Crohn's, ulcerative colitis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2005-04; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Srikala Sridhar, Principal Investigator — Princess Margaret Hospital Phase 2 Consortium
Locations (1):
- Princess Margaret Hospital Phase 2 Consortium, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Sorafenib Tosylate): Patients receive oral sorafenib twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  sorafenib tosylate: Given orally
  laboratory biomarker analysis: Correlative studies
Period: Overall Study
Arm/Group | Treatment (Sorafenib Tosylate)
Started | 17
Completed | 17
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All participants
Arm/Group | Treatment (Sorafenib Tosylate)
Number analyzed (Participants) | 17
Age, Continuous [Median (Full Range); unit: years] | 67 [40 to 85]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 14
Region of Enrollment [Number; unit: participants]
  Canada | 17

OUTCOME MEASURES:

1. Primary Outcome: Number of Paricipants With Tumour Response Defined as Partial or Complete Response Per the RECIST 1.0 Criteria
Description: Per Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), disappearance of all target lesions; Partial Response (PR), at least 30% decrease in the sum of the longest diameter of target lesions; Objective Response (OR) = CR + PR.
Time Frame: Up to 5 years
Measure: Number; unit: participants
Arm/Group | Treatment (Sorafenib Tosylate)
Number analyzed (Participants) | 17
participants | 0

2. Secondary Outcome: Number of Participants With Stable Disease for More Than 3 Months
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD), >=20% increase in the sum of the longest diameter of target lesions; Stable Disease (SD), neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
Time Frame: From the start of the treatment until the criteria for progression are met, up to 5 years
Population: Stable disease for more than 3 months
Measure: Number; unit: participants
Arm/Group | Treatment (Sorafenib Tosylate)
Number analyzed (Participants) | 17
participants | 1

3. Secondary Outcome: Time to Progression
Description: Progression is defined using the Response Evaluation Criteria In Solid Tumours Criteria (RECIST v1.0) as at least a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in non-target lesions, or the appearance of new lesions.
Time Frame: Up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Sorafenib Tosylate)
Number analyzed (Participants) | 17
months | 1.9 [1.7 to 4.3]

4. Secondary Outcome: Progression-free Survival
Description: Summary statistics, such as the mean, median, counts and proportion, will be used to summarize the patients. Survival estimates will be computed using the Kaplan-Meier method. Potential association between variables will be measured using Pearson correlation coefficients, chi-square tests, one- or two-sample t-tests or logistic regression analyses as appropriate. Non-parametric tests such as Spearman correlation coefficients, Fisher's exact tests and Wilcoxon tests may be substituted if necessary. 95% confidence intervals will be constructed and selected results will be illustrated.
Time Frame: From start of treatment to progression or death, assessed up to 1 year
Population: 3 months progression free survival
Measure: Median (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Sorafenib Tosylate)
Number analyzed (Participants) | 14
percentage of participants | 27 [12 to 61]

5. Secondary Outcome: Frequency of Common Grade 3 Adverse Events
Description: Will be tabulated using counts and proportions detailing frequently occurring, serious and severe events of interest.
Time Frame: Up to 5 years
Measure: Number; unit: common grade 3 events
Arm/Group | Treatment (Sorafenib Tosylate)
Number analyzed (Participants) | 17
common grade 3 events | 3

ADVERSE EVENTS:
Arm/Group | Treatment (Sorafenib Tosylate)
Serious Adverse Events (participants affected / at risk) | 2/17
Other Adverse Events (participants affected / at risk) | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Sorafenib Tosylate) (N=17)
Multi-organ failure (General disorders) | 1 (1)
Death NOS (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Sorafenib Tosylate) (N=17)
Fatigue (General disorders) | 16 (16)
Anorexia (Metabolism and nutrition disorders) | 12 (12)
Constipation (Gastrointestinal disorders) | 11 (11)
Abdominal pain (Gastrointestinal disorders) | 11 (11)
Abdominal pain (Gastrointestinal disorders) | 4 (4)
back pain (Musculoskeletal and connective tissue disorders) | 4 (4)
hand-foot reaction (Skin and subcutaneous tissue disorders) | 3 (3)
bladder infection (Infections and infestations) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less